CLINICAL TRIAL: NCT00484315
Title: A Prospective Evaluation in a Randomized Trial of the Safety and Efficacy of the Use of the TAXUS Element Paclitaxel-Eluting Coronary Stent System for the Treatment of De Novo Coronary Artery Lesions
Brief Title: TAXUS PERSEUS Workhorse
Acronym: PERSEUS WH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2037; S2037-PIVOT-2006
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Results first posted 2011-06-28 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Disease
Keywords: drug-eluting stent; paclitaxel-eluting stent; DES
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAXUS Element (Experimental)
  Interventions: Device: Percutaneous coronary intervention (PCI) with paclitaxel-eluting stent (TAXUS Element) implantation
- TAXUS Express (Active Comparator)
  Interventions: Device: Percutaneous coronary intervention (PCI) with paclitaxel-eluting stent (TAXUS Express) placement

INTERVENTIONS:
Device: Percutaneous coronary intervention (PCI) with paclitaxel-eluting stent (TAXUS Element) implantation — TAXUS Element stent placement
  Arms: TAXUS Element
Device: Percutaneous coronary intervention (PCI) with paclitaxel-eluting stent (TAXUS Express) placement — TAXUS Express Stent Implant
  Arms: TAXUS Express

SUMMARY:
The purpose of the TAXUS PERSEUS Workhorse trial is to evaluate the safety and efficacy of the next-generation Boston Scientific TAXUS paclitaxel-eluting coronary stent system (TAXUS® ElementTM) for the treatment of de novo atherosclerotic lesions of up to 28 mm in length in native coronary arteries of 2.75 mm to 4.0 mm diameter.

DETAILED DESCRIPTION:
This is a prospective, 3:1 randomization, multi-center trial to assess the TAXUS® Element™ Paclitaxel-Eluting Coronary Stent System for the treatment of de novo atherosclerotic lesions of up to 28 mm in length in native coronary arteries ≥ 2.75 mm and ≤ 4.0 mm in diameter, compared to a control group of TAXUS Express2 Paclitaxel-Eluting Coronary Stent System .

One thousand two hundred sixty-four (1264) subjects will be treated with either the TAXUS® Element™ stent or the TAXUS® Express2 ™stent at a maximum of 100 clinical sites. Randomization to treatment group will be unbalanced 3:1 towards the test group to gain maximum clinical experience with the new TAXUS® Element™ platform. Follow-up at 30 days, 9 months and 12 months will be completed in all subjects enrolled in the study. Angiographic follow-up at 9 months will be completed in a subset of three hundred thirty (330) subjects enrolled in the study. Subjects will be randomly allocated to the angiographic subset at participating sites through the Interactive Voice Response System (IVRS).

Eligible subjects will have annual follow-up until 5 years post-index procedure.

ELIGIBILITY:
Clinical Inclusion Criteria:

* Subject is ≥ 18 years old
* Eligible for percutaneous coronary intervention (PCI)
* Documented stable angina pectoris (Canadian Cardiovascular Society [CCS] Classification 1, 2, 3, or 4) or unstable angina pectoris (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia
* Acceptable candidate for coronary artery bypass grafting (CABG)
* Left ventricular ejection fraction (LVEF) is ≥ 30%
* Subject (or legal guardian) understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed
* Subject willing to comply with all specified follow-up evaluations

Clinical Exclusion Criteria:

* Contraindication to aspirin (ASA), or to both clopidogrel and ticlopidine
* Known hypersensitivity to paclitaxel
* Known allergy to stainless steel
* Known allergy to platinum
* Previous treatment of the target vessel with any anti-restenotic drug-coated or drug-eluting coronary stent
* Previous treatment of the target vessel with a bare metal stent (BMS) within 9 months of the index procedure
* Previous treatment of any non-target vessel with any anti-restenotic drug-coated or drug-eluting coronary stent within 9 months of the index procedure
* Previous treatment with intravascular brachytherapy in the target vessel
* Planned PCI or CABG post-index procedure
* Planned or actual target vessel treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon or transluminal extraction catheter immediately prior to stent placement
* Myocardial infarction (MI) within 72 hours prior to index procedure
* Cerebrovascular accident (CVA) within the past 6 months
* Cardiogenic shock
* Acute or chronic renal dysfunction
* Prior anaphylactic reaction to contrast agents
* Leukopenia
* Thrombocytopenia
* Thrombocytosis
* Active peptic ulcer or active gastrointestinal (GI) bleeding
* Current treatment, or past-treatment within 12-months of the index procedure, with paclitaxel or other chemotherapeutic agents
* Anticipated treatment with paclitaxel or oral rapamycin during any period in the 9-months after the index procedure
* Known intention to procreate within 9 months after the index procedure
* Positive pregnancy test within 7 days before the index procedure, or lactating
* Life expectancy of less than 24 months due to other medical conditions
* Co-morbid condition(s) that could limit subject's ability to comply with study follow-up requirements or impact study scientific integrity
* Currently participating in another investigational drug or device study

Angiographic Inclusion Criteria:

* Target Lesion

  * Target lesion located in native coronary artery
  * Target lesion must be de novo
  * Target lesion diameter stenosis ≥ 50%
  * Reference vessel diameter (RVD) ≥ 2.75 mm to ≤ 4.0 mm
  * Cumulative target lesion length ≤ 28 mm (area to be treated may be composed of multiple lesions but must be completely coverable by one study stent)
  * Target lesion is successfully pre-dilated
* One non-target lesion may be treated in a non-target vessel as follows:

  * Non-target lesion in non-target vessel must be treated with commercially available TAXUS stent if use of drug eluting stent required
  * Treatment must be deemed a clinical angiographic success, without requiring use of unplanned additional stents(s)
  * Treatment must be completed prior to treatment of target vessel

Angiographic Exclusion Criteria

* Target lesion located in left main artery, whether protected or unprotected
* Target lesion is a chronic total occlusion (TIMI flow ≤ 1)
* Target lesion is restenotic
* Target lesion is located in a saphenous vein graft or mammary artery graft
* Target lesion is accessed via saphenous vein graft or mammary artery graft
* Target lesion is < 5 mm from bare metal stent (BMS)
* Target lesion < 5 mm from ostium
* Target lesion < 5 mm from side branch vessel ≥ 2.0 mm in diameter (Exceptions: subject may be enrolled if side branch is 100% occluded or if side branch is protected with a patent graft)
* Untreated lesions with ≥ 50% diameter stenosis or thought to impair flow remaining in target vessel at a location with ≥ 2.0mm RVD
* Target lesion and/or target vessel proximal to target lesion moderately or severely calcified
* Target lesion and/or target vessel proximal to target lesion severely tortuous
* Target lesion located within or distal to a > 60° bend in target vessel
* Target vessel with angiographic presence of probable or definite thrombus
* Unprotected left main coronary artery disease
* Protected left main coronary artery disease with target lesion in Left Anterior Descending artery (LAD) or Left Circumflex artery (LCx). Subject may be enrolled if only lesion is target lesion in Right Coronary Artery (RCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1264 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean J Kereiakes, MD, Principal Investigator — The Christ Hospital; Louis A Cannon, MD, Principal Investigator — Cardiac and Vascular Research Center of Northern Michigan
Locations (90):
- United States (82):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Medical Center East, Birmingham, Alabama
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Alvarado Hospital, La Jolla, California
  - Scripps Clinic, La Jolla, California
  - Scripps Memorial Hospital, La Jolla, California
  - University of California, Davis Medical Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Mediquest Research at Munroe Regional Medical Center, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Kaiser Foundation Hospitals, Honolulu, Hawaii
  - Evanston Northwestern, Evanston, Illinois
  - St. Anthony's Medical Center, Rockford, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Northern Indiana Research Alliance / Lutheran Hospital of Indiana, Fort Wayne, Indiana
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - St. Vincent's Hospital, Indianapolis, Indiana
  - Trinity Terrace Park, Davenport, Iowa
  - Iowa Heart Center, Des Moines, Iowa
  - Maine Medical Center, Portland, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Lakeland Hospitals at St. Joseph, Saint Joseph, Michigan
  - St. Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mercy Hospital, Minneapolis, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Anthony's Medical Center, St Louis, Missouri
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Heart Hospital of New Mexico, Albuquerque, New Mexico
  - St. Joseph's Hospital Health Center, Liverpool, New York
  - Lenox Hill Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Main Line Health Heart Center, Bryn Mawr, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Sisters of Charity Providence Hospital, Columbia, South Carolina
  - University Medical Center-Greenville Memorial Hospital, Greenville, South Carolina
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - Methodist DeBakey Heart Center, Houston, Texas
  - TexSAn Heart Hospital, San Antonio, Texas
  - Trinity Mother Frances Health System, Tyler, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Lynchburg General Hospital, Lynchburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - St. Mary's Medical Center, Huntington, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - CaRE Foundation, Inc., Wausau, Wisconsin
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, SA, Australia, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincents Public,, Fitzroy, Victoria
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington
- National Heart Centre, Singapore, Singapore

REFERENCES:
- [Derived] Kereiakes DJ, Cannon LA, Feldman RL, Popma JJ, Magorien R, Whitbourn R, Dauber IM, Rabinowitz AC, Ball MW, Bertolet B, Kabour A, Foster MC, Wang JC, Underwood P, Dawkins KD. Clinical and angiographic outcomes after treatment of de novo coronary stenoses with a novel platinum chromium thin-strut stent: primary results of the PERSEUS (Prospective Evaluation in a Randomized Trial of the Safety and Efficacy of the Use of the TAXUS Element Paclitaxel-Eluting Coronary Stent System) trial. J Am Coll Cardiol. 2010 Jul 20;56(4):264-71. doi: 10.1016/j.jacc.2010.04.011. Epub 2010 May 20. PMID 20493653
- [Derived] Allocco DJ, Cannon LA, Britt A, Heil JE, Nersesov A, Wehrenberg S, Dawkins KD, Kereiakes DJ. A prospective evaluation of the safety and efficacy of the TAXUS Element paclitaxel-eluting coronary stent system for the treatment of de novo coronary artery lesions: design and statistical methods of the PERSEUS clinical program. Trials. 2010 Jan 7;11:1. doi: 10.1186/1745-6215-11-1. PMID 20059766

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of 1264 subjects was planned; 1262 (942 TAXUS Element and 320 TAXUS Express) were enrolled and randomized at 90 centers by October 1, 2008. A total of 330 subjects were randomly assigned to protocol-mandated 9-month angiographic follow-up (angiographic subset).
Groups:
- TAXUS Element: Participants randomized to treatment with TAXUS Element paclitaxel-eluting stent (investigational device)
- TAXUS Express: Participants randomized to treatment with TAXUS Express paclitaxel-eluting stent (control device)
Period: 12-Month Clinical Follow-up
Arm/Group | TAXUS Element | TAXUS Express
Started | 942 | 320
Completed | 914 | 311
Not Completed | 28 | 9
Not completed — Death | 6 | 2
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Missed 12-Month Visit | 13 | 4
Not completed — Withdrawn at Investigator's discretion | 3 | 2
Period: 9-Month Angiographic Follow-up
Arm/Group | TAXUS Element | TAXUS Express
Started | 256 | 74
Completed | 228 | 61
Not Completed | 28 | 13
Not completed — No 9-Month Angiography Performed | 25 | 11
Not completed — Not Evaluable for Angiography Analysis | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAXUS Element | TAXUS Express | Total
Number analyzed (Participants) | 942 | 320 | 1262
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 540 | 163 | 703
  >=65 years | 402 | 157 | 559
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.6) | 63.5 (9.5) | 62.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 100 | 375
  Male | 667 | 220 | 887
Race/Ethnicity, Customized [Number; unit: participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Hispanic or Latino | 10 | 6 | 16
    Caucasian | 872 | 296 | 1168
    Asian | 15 | 6 | 21
    Black of African heritage | 37 | 13 | 50
    Native Hawaiian or other Pacific Islander | 4 | 1 | 5
    American Indian or Alaska native | 3 | 0 | 3
    Other | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 859 | 290 | 1149
  Singapore | 6 | 2 | 8
  Australia | 60 | 22 | 82
  New Zealand | 17 | 6 | 23
Cardiac History [Number; unit: participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Previous Percutaneous Coronary Intervention (PCI) | 216 | 80 | 296
    Previous Coronary Artery Bypass Graft (CABG) | 42 | 20 | 62
    Previous Myocardial Infarction (MI) | 195 | 60 | 255
    Congestive Heart Failure | 56 | 24 | 80
    Stable Angina | 629 | 213 | 842
    Unstable Angina | 195 | 68 | 263
    Silent Ischemia | 117 | 39 | 156
Cardiac History: Ejection Fraction [Mean (Standard Deviation); unit: ejection fraction percent] | 58.0 (9.3) | 57.8 (9.8) | 57.9 (9.4)
Cardiac Risk Factors [Number; unit: participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Smoking, Ever | 611 | 216 | 827
    Medically Treated Diabetes | 232 | 80 | 312
    Hyperlipidemia Requiring Medication | 717 | 243 | 960
    Hypertension Requiring Medication | 709 | 256 | 965
    Family History of Coronary Artery Disease | 589 | 196 | 785
Comorbidities [Number; unit: participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Peripheral Vascular Disease | 99 | 36 | 135
    History of Transient Ischemic Attack | 30 | 14 | 44
    History of Cerebrovascular Accident | 30 | 12 | 42
    History of Renal Disease | 45 | 11 | 56
    History of Gastrointestinal Bleeding | 9 | 7 | 16
Lesion Characteristic: Target Lesion Vessel [Number; unit: participants]
  Left Anterior Descending Artery | 406 | 140 | 546
  Left Circumflex Artery | 217 | 69 | 286
  Right Coronary Artery | 319 | 111 | 430
Lesion Characteristic: Lesion Location [Number; unit: participants]
  Ostial | 25 | 8 | 33
  Proximal | 368 | 128 | 496
  Mid | 485 | 154 | 639
  Distal | 64 | 30 | 94
Lesion Characteristics [Mean (Standard Deviation); unit: millimeter]
  Reference Vessel Diameter | 2.8 (0.5) | 2.8 (0.5) | 2.8 (0.5)
  Minimum Lumen Diameter | 0.8 (0.3) | 0.8 (0.4) | 0.8 (0.3)
  Lesion Length | 14.2 (6.1) | 14.1 (5.8) | 14.2 (6.0)
  Sidebranch Stenosis | 24.4 (28.1) | 25.7 (28.8) | 24.7 (28.3)
Lesion Characteristic: Percent Diameter Stenosis [Mean (Standard Deviation); unit: percent] | 72.1 (10.9) | 71.7 (10.9) | 72.0 (10.9)
Lesion Characteristics [Number; unit: participants] — The same participant may be included in more than one category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    Eccentric Lesion | 487 | 161 | 648
    > 45 Degree Bend | 61 | 22 | 83
    > 90 Degree Bend | 2 | 1 | 3
    Tortuosity, any | 59 | 14 | 73
    Calcification, any | 228 | 86 | 314
    Total Occlusion | 6 | 2 | 8
    Bifurcation | 343 | 129 | 472
Lesion Characteristics: American College of Cardiology (ACC)/American Heart Association (AHA) Class [Number; unit: participants] — Type A lesions: minimally complex, readily accessible, non angulated, smooth contour, little to no calcification, less than totally occlusive, not ostial in location, no major side branch involvement, and an absense of thrombus.
  Type B lesions: moderately complex, eccentric, moderate tortuosity and angulation, moderate or heavy calcification, total occlusion < 3 months old, ostial in location, with presence of thrombus.
  Type C lesions: severely complex, diffuse, excessive tortuosity and angulation, total occlusions > 3 months old, degenerated vein grafts and friable lesions.
  participants
    Type A | 79 | 28 | 107
    Type B1 | 233 | 85 | 318
    Type B2 | 384 | 130 | 514
    Type C | 246 | 77 | 323
Lesion Characteristic - Pre-Procedure Thrombolysis In Myocardial Infarction (TIMI) Flow [Number; unit: participants] — TIMI 0 - No perfusion TIMI 1 - Penetration with minimal perfusion TIMI 2 - Partial perfusion TIMI 3 - Complete perfusion
  participants
    TIMI 0 | 2 | 2 | 4
    TIMI 1 | 4 | 0 | 4
    TIMI 2 | 34 | 4 | 38
    TIMI 3 | 902 | 314 | 1216

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure (TLF) at 12 Months Post-index Procedure. TLF is Defined as Any Ischemia-driven Revascularization of the Target Lesion, Myocardial Infarction (Q-wave and Non-Q-wave), or Death Related to the Target Vessel.
Description: The number of participants who experience a TLF through 365 days post-procedure out of the participants who have either had a TLF within 365 days post-procedure or who were TLF-free with last follow-up at least 335 days post-procedure.
Time Frame: 12 months post-index procedure
Population: The primary analysis set for the non-inferiority testing of the primary endpoint, 12-month TLF, is the per protocol analysis set. All randomized participants who had the randomly assigned study stent implanted in the target coronary artery are included.
Measure: Number; unit: participants
Groups:
- TAXUS Element; TAXUS Express: Paclitaxel-eluting stent (PES) implanted using standard percutaneous coronary intervention (PCI) technique
Arm/Group | TAXUS Element | TAXUS Express
Number analyzed (Participants) | 915 | 309
participants | 51 | 19
Statistical Analysis 1: Comparison: TAXUS Element vs TAXUS Express; Bayesian modeling was used to determine if the 12-month TLF rate for the TAXUS Element stent was non-inferior to the 12-month TLF rate in the TAXUS Express2 control. The null hypothesis was that the TAXUS Element TLF rate is at least 4.1% greater than the TAXUS Express TLF rate. The alternative hypothesis was that the TAXUS Element TLF rate is less than 4.1% greater than the TAXUS Express TLF rate; Test type: Non-Inferiority or Equivalence — Non-inferiority of the TAXUS Element stent was to be accepted if the Bayesian posterior probability that the difference in 12-month TLF between TAXUS Element and TAXUS Express was < 4.1%, given the data, was at least 95%. The sample size of 1264 subjects (resulting in 1200 after accounting for 5% attrition) was determined through simulations based on Bayesian modeling; p = 0.9996, Bayesian modeling — The p-value is the posterior probability that the difference in 12-month TLF between TAXUS Element and TAXUS Express was < 4.1%, given the data observed; Median Difference (Final Values) = -0.570, 95% CI 1-sided [upper limit 1.85], Standard Deviation 0.0155 — Values are based on the posterior distribution of the difference in TLF rates between TAXUS Element and TAXUS Express. The upper limit is the 1-Sided 95% posterior credible interval, based off the 95th percentile of the posterior distribution

2. Secondary Outcome: In-segment Percent Diameter Stenosis at 9 Months Post-index Procedure
Description: The minimum lumen diameter in the analysis segment at 9-months post-index procedure, divided by the reference vessel diameter at baseline. The analysis segment ("in-segment") is defined as the proximal edge, stented area, and the distal edge, where each edge segment contains up to 5mm immediately outside the stent.
Time Frame: 9 months post-index procedure
Population: All patients from the per protocol analysis set who were randomized to the angiographic subset and completed their angiographic follow-up were analyzed for the secondary endpoint.
Measure: Mean (Standard Deviation); unit: percent diameter stenosis
Arm/Group | TAXUS Element | TAXUS Express
Number analyzed (Participants) | 228 | 60
percent diameter stenosis | 26.1 (17.71) | 26.28 (17.6)
Statistical Analysis 1: Comparison: TAXUS Element vs TAXUS Express; Natural log (ln) transformation was used to improve normality of the secondary endpoint distribution. Bayesian modeling was used to determine if the mean ln(9-month percent diameter stenosis) for the TAXUS Element stent was non-inferior to the mean ln(9-month %DS) for TAXUS Express. Null hypothesis was that the TAXUS Element mean was at least 0.20 greater than the TAXUS Express mean. Alternative hypothesis was that the TAXUS Element mean is less than 0.20 greater than the TAXUS Express TLF mean; Test type: Non-Inferiority or Equivalence — Non-inferiority of the TAXUS Element stent was to be accepted if the Bayesian posterior probability that the difference in mean ln(9-month percent diameter stenosis) between TAXUS Element and TAXUS Express was < 0.20, given the data, was at least 95%. The sample size of 330 subjects (resulting in 280 after accounting for 15% attrition) was determined through simulations based on Bayesian modeling; p = 0.9970, Bayesian modeling — P-value is posterior probability that the difference in mean ln(9-month percent diameter stenosis) between TAXUS Element and TAXUS Express was < 0.20, given the data observed. Non-inferiority was concluded, as this probability is greater than 95%; Mean Difference (Final Values) = -0.0294, 95% CI 1-sided [upper limit 0.1078], Standard Deviation 0.08253 — Based on posterior distribution of the difference in mean ln(9-month percent diameter stenosis) between TAXUS Element and TAXUS Express. Upper limit is 1-Sided 95% posterior credible interval, based off the 95th percentile of posterior distribution

ADVERSE EVENTS:
Time Frame: Site reported serious and non-serious adverse events were collected through 365 days.
Arm/Group | TAXUS Element | TAXUS Express
Serious Adverse Events (participants affected / at risk) | 334/942 | 110/320
Other Adverse Events (participants affected / at risk) | 277/942 | 97/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAXUS Element (N=942) | TAXUS Express (N=320)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 73 (84) | 27 (28)
Angina unstable (Cardiac disorders) | 18 (19) | 6 (7)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 14 (16) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (4) | 2 (2)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 4 (5) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 7 (8) | 5 (9)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 9 (9) | 3 (3)
Coronary artery dissection (Cardiac disorders) | 10 (10) | 10 (10)
Coronary artery embolism (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 18 (19) | 5 (5)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 24 (24) | 5 (5)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 6 (6) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular asystole (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 3 (5) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (6) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Splenic artery aneurysm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Catheter site haematoma (General disorders) | 4 (4) | 3 (3)
Catheter site haemorrhage (General disorders) | 4 (4) | 2 (2)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 53 (61) | 15 (18)
Pain (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 4 (6)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 3 (4)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (9) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 3 (3) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 4 (5) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 3 (4)
Mental status changes (Psychiatric disorders) | 4 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3)
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (3) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Intermittent claudication (Vascular disorders) | 10 (11) | 0 (0)
Myocardial infarction (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 4 (5) | 4 (4)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 7 (7) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAXUS Element (N=942) | TAXUS Express (N=320)
Angina pectoris (Cardiac disorders) | 98 (114) | 40 (44)
Catheter site haematoma (General disorders) | 46 (47) | 19 (22)
Catheter site haemorrhage (General disorders) | 28 (28) | 16 (18)
Non-cardiac chest pain (General disorders) | 120 (150) | 32 (36)
Back pain (Musculoskeletal and connective tissue disorders) | 55 (56) | 18 (19)

LIMITATIONS AND CAVEATS:
The comparator control for PERSEUS Workhorse study was chosen based on commercially available stent (TAXUS Express) at the time of study enrollment. Thus, the comparator group does not represent the most recently available paclitaxel-eluting stent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall have the right to publish the results, provided that before publishing, the PI shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.